CLINICAL TRIAL: NCT00269308
Title: Randomized Clinical Trial of Chiropractic Manual Therapy Plus Home Exercise, Supervised Exercise Plus Home Exercise and Home Exercise Alone For Individual 65 and Over With Chronic Mechanical Neck Pain
Brief Title: Chiropractic and Exercise for Seniors With Neck Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern Health Sciences University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Berman Center for Outcomes and Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18HP01425
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Neck Pain
Keywords: Randomized; Clinical Trial; Neck Pain; Chiropractic; Manual Therapies; Exercise
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- 1 (Experimental): Chiropractic Manual Treatment + Home Exercise
  Interventions: Procedure: Chiropractic Manual treatment + home exercise ( procedure+behavior)
- 2 (Experimental): Supervised Rehabilitative Exercise + Home Exercise
  Interventions: Procedure: Supervised rehabilitative exercise + home exercise
- 3 (Active Comparator): Home Exercise
  Interventions: Behavioral: Home exercise

INTERVENTIONS:
Procedure: Chiropractic Manual treatment + home exercise ( procedure+behavior) — The number of treatments will be determined by the individual chiropractor. Chiropractic manual treatment will be limited to gentle spinal manipulation and mobilization with light soft tissue massage as indicated to facilitate the manual therapy.
  Patients will attend 4, 1-hour small-group sessions at weeks 1, 2, 4 and 8. At the first two sessions they will be given information about neck pain and shown exercises to perform at home. Emphasis will be placed on the importance of staying active
  Arms: 1
Procedure: Supervised rehabilitative exercise + home exercise — The rehabilitative exercise program will consist of 20, 1 hour small-group sessions. It is a modification of exercise protocols used in previous studies by the investigators and others and incorporates recommendations of leading rehabilitative exercise specialists. The program will include exercises that reduce joint stiffness and relax elastic structures resulting in lower joint loads during movements.
  Patients will attend 4, 1-hour small-group sessions at weeks 1, 2, 4 and 8. At the first two sessions they will be given information about neck pain and shown exercises to perform at home. Emphasis will be placed on the importance of staying active
  Arms: 2
Behavioral: Home exercise — Patients will attend 4, 1-hour small-group sessions at weeks 1, 2, 4 and 8. At the first two sessions they will be given information about neck pain and shown exercises to perform at home. Emphasis will be placed on the importance of staying active.
  Arms: 3

SUMMARY:
The purpose of this randomized clinical trial is to assess the relative effectiveness of three conservative treatment approaches for seniors with chronic neck pain: 1) chiropractic manual treatment plus home exercise, 2) supervised exercise plus home exercise and 3) home exercise alone.

DETAILED DESCRIPTION:
Neck pain (NP) is a considerable health problem, affecting both young and elderly individuals. Of particular concern is the negative impact NP may have on the functional ability of the geriatric population, already challenged by decreased mobility and balance associated with ageing. Chiropractic manual treatment and rehabilitative exercise have demonstrated potential for the treatment of NP in younger individuals, but have yet to be rigorously tested in the elderly.

The broad, long-term objective of this research is to identify effective therapies for patients, 65 years and older, who suffer with chronic neck pain and to enhance their functional capacity.

Primary Aims

• To determine the relative clinical effectiveness of 1) chiropractic manual treatment and home exercise, 2) supervised rehabilitative exercise and home exercise, and 3) home exercise alone in both the short-term (after 12 weeks) and long-term (after 52 weeks), using patient-rated neck pain as the main outcome measure.

Secondary Aims

* To estimate the short- and long-term relative effectiveness of the three interventions using:

  * Patient-rated outcomes: neck related disability, general health status, patient satisfaction, improvement, and medication use measured by self-report questionnaires;
  * Objective functional performance outcomes: neck motion, strength and endurance, and functional ability measured by examiners masked to treatment group assignment;
  * Cost measures: direct and indirect costs, and cost utility of treatment measured by questionnaires, phone interviews, and medical records.
* To describe patients' perceptions of treatment and the issues they consider when determining their satisfaction with care.

This project is a collective effort by a multidisciplinary team, with an established record of collaborative research in the area of neck and back pain. The results of this study will provide valuable information for elderly neck pain sufferers and the clinicians who treat them.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain (Defined as current episode more than 12 weeks duration.)
* Quebec Task Force classifications 1, 2, 3 and 4. This includes patients with neck pain, stiffness or tenderness, with or without musculoskeletal and neurological signs.
* 65 years of age and older
* Independent ambulation
* Community dwelling (residency outside nursing home)
* Score of 20 or more on Folstein Mini-Mental State Examination
* Stable prescription medication plan (no changes in prescription medications that affect musculoskeletal pain in previous month)

Exclusion Criteria:

* Referred neck pain from local joint lesions of the upper extremities or from visceral diseases
* Significant infectious disease
* Ongoing treatment for neck pain by other health care providers
* Mean neck pain score of less than 20 percentage points
* Contraindications to exercise Determined by history or by referral to supplementary diagnostic tests (i.e., uncontrolled arrhythmias, third degree heart block, recent ECG changes, unstable angina, acute myocardial infarction, acute congestive heart failure, cardiomyopathy, valvular heart disease, poorly controlled blood pressure, uncontrolled metabolic disease)
* Contraindications to spinal manipulation (i.e. Progressive neurological deficits, blood clotting disorders, severe osteoporosis, infectious and non-infectious inflammatory or destructive tissue changes of the spine)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 241 (Actual)
Dates: Start 2003-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Patient-rated pain (0-10 scale, 11 box) | short term = 12 weeks; long term = 52 weeks

SECONDARY OUTCOMES:
General Health | short term = 12 weeks; long term = 52 weeks
Disability | short term = 12 weeks; long term = 52 weeks
Improvement | short term = 12 weeks; long term = 52 weeks
Satisfaction | short term = 12 weeks; long term = 52 weeks
Medication use | short term = 12 weeks; long term = 52 weeks
Biomechanical tests: Cervical spine motion, Strength and Endurance, Functional Ability, Observed Pain Behavior | short term = 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gert Bronfort, DC, PhD, Principal Investigator — Northwestern Health Sciences University
Locations (1):
- Wolfe-Harris Center for Clinical Studies, Northwestern Health Sciences University, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Leininger B, McDonough C, Evans R, Tosteson T, Tosteson AN, Bronfort G. Cost-effectiveness of spinal manipulative therapy, supervised exercise, and home exercise for older adults with chronic neck pain. Spine J. 2016 Nov;16(11):1292-1304. doi: 10.1016/j.spinee.2016.06.014. Epub 2016 Jun 23. PMID 27345747
- [Derived] Maiers M, Bronfort G, Evans R, Hartvigsen J, Svendsen K, Bracha Y, Schulz C, Schulz K, Grimm R. Spinal manipulative therapy and exercise for seniors with chronic neck pain. Spine J. 2014 Sep 1;14(9):1879-89. doi: 10.1016/j.spinee.2013.10.035. Epub 2013 Nov 10. PMID 24225010
- [Derived] Maiers MJ, Hartvigsen J, Schulz C, Schulz K, Evans RL, Bronfort G. Chiropractic and exercise for seniors with low back pain or neck pain: the design of two randomized clinical trials. BMC Musculoskelet Disord. 2007 Sep 18;8:94. doi: 10.1186/1471-2474-8-94. PMID 17877825
- See also: Related Info — http://www.nwhealth.edu/research/WHCCS/